CLINICAL TRIAL: NCT05184257
Title: The Effectiveness of Zoladex® 10.8 mg Compared to Zoladex® 3.6mg in the Treatment of Premenopausal and Perimenopausal Hormone Receptor Positive Breast Cancer: A Real-World Study
Brief Title: Zoladex® 10.8 BC RWS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8664R00002
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Drugs: The study drug is Zoladex® 10.8 mg. The maximum observation time window for effectiveness analysis is 28 (24+4) weeks.
- Comparison Drugs: The comparison drug is Zoladex® 3.6 mg. The maximum observation time window for effectiveness analysis is 28 (24+4) weeks.

SUMMARY:
This is a multi-center, retrospective-prospective, observational, active-control, non-inferiority, real world study using hospital medical record data, with objectives to evaluate E2 suppressive effect of Zoladex® 10.8 mg is non-inferior to Zoladex® 3.6 mg. Eligible breast cancer patients who received Zoladex® from January 1st, 2015 till December 31st, 2021(including December 31st, 2021) will be identified and included for retrospective data collection and analyses in this study. And prospective data will be monthly collected of eligible patients receiving Zoladex® after January 1st, 2022 (including January 1st, 2022) until approximately 1000 patients being included in this study for analysis. (If site has specific identification of retrospective data and prospective data, it will be subject to the requirement of site). The first date of the presence of Zoladex® treatment or prescription record for breast cancer during the study period will be considered the index date for patients. According to the Zoladex® treatment at the index date, patients will be categorized into two cohorts: Zoladex® 10.8 mg or Zoladex® 3.6 mg.

About 10-15 hospitals will be included in this study. To be considered, the hospitals need to have relatively large number of eligible patients, geographic representativeness and willingness to participate in this study. Approximately 1000 eligible patients from selected hospitals during the study period will be included and matched with propensity scores. It is expected that at least 150 matched patients in each of the two cohorts will eventually be included in the primary endpoint analysis. The final subject number will be based on the actual situation of the study.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with primary breast cancer
* Female, ≥18 years old (at index date)
* HR positive
* Receive Zoladex® 10.8 mg or Zoladex® 3.6 mg treatment
* Premenopausal status prior to the treatment of Zoladex®. Baseline premenopausal status will be confirmed if the patient's last E2 measurement within 180 days prior to the index date indicated premenopausal status or there was a recorded menstrual history within 180 days prior to the index date
* At least one actual or expected E2 testing measurement within 8-28 weeks of the index date Exclusion Criteria
* Patients received concurrent treatments that may affect E2 testing results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with premenopausal and perimenopausal breast cancer
Sampling Method: Probability Sample
Enrollment: 1176 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with serum E2 suppression at 12 weeks (±4 weeks). Serum E2 suppression is defined as an E2 value below the upper limit of the menopausal reference range | serum E2 suppression at 12 weeks (±4 weeks) after Zoladex® treatment
  To assess the E2 suppressive effect of Zoladex® 10.8 mg is non-inferior to Zoladex® 3.6 mg at 12th week for the treatment of patients with premenopausal and perimenopausal breast cancer.

SECONDARY OUTCOMES:
Proportion of patients with serum E2 suppression at 24 weeks (±4 weeks). Serum E2 suppression was defined as an E2 value below the upper limit of the menopausal reference range | serum E2 suppression at 24 weeks (±4 weeks) after Zoladex®
  To assess the E2 suppressive effect of Zoladex® 10.8 mg and Zoladex® 3.6 mg at 24th week for the treatment of patients with premenopausal and perimenopausal breast cancer

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangan
  - Research Site, Guangyuan
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Nantong
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Xining

REFERENCES:
- [Derived] Wang Y, Wang X, Wu J, Liu H, Zhao J, Huang J, Liu J, Gong Y, Wang H, Yang H, Zou G, Ouyang Q, Jiang G, Liu H, Ni S, Xu B, Yu J. Real-world effectiveness of goserelin 10.8-mg compared to goserelin 3.6-mg in premenopausal and perimenopausal Chinese patients with hormone receptor positive breast cancer: a cohort study. J Natl Cancer Cent. 2025 May 20;5(4):392-401. doi: 10.1016/j.jncc.2025.02.006. eCollection 2025 Aug. PMID 40814439
- See also: CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8664R00002&attachmentIdentifier=45ff70bd-03ba-4deb-bd28-0891932e706f&fileName=D8664R00002-redacted_CSR_synopsis.pdf&versionIdentifier=